CLINICAL TRIAL: NCT04980417
Title: Concomitant Cholecystectomy With Bariatric Surgery Versus Delayed Post Bariatric Cholecystectomy for Obesity With Gallstone
Brief Title: Concomitant Versus Delayed Cholecystectomy for Management of Obesity With Gallstone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor & consultant of general surgery, Department of Surgery, Minia university hospital, Egypt, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fac.med 21.32
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Morbid Obesity; Gallstone
MeSH Terms: conditions — Obesity, Morbid; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concomitant cholecystectomy (Experimental): concomitant cholecystectomy with bariatric procedure
  Interventions: Procedure: concomitant cholecystectomy
- delayed cholecystectomy (Active Comparator): delayed cholecystectomy
  Interventions: Procedure: concomitant cholecystectomy

INTERVENTIONS:
Procedure: concomitant cholecystectomy — delayed cholecystectomy
  Other Names: delayed cholecystectomy

SUMMARY:
in this study we compare the results of concomitant cholecystectomy with bariatric surgery versus delayed cholecystectomy for management of gallstone in obese patients

DETAILED DESCRIPTION:
in this study we compare the results of concomitant cholecystectomy with bariatric surgery versus delayed cholecystectomy for management of gallstone in obese patients. patients will be divided into 2 group: group1, will be operated by the bariatric surgery and cholecystectomy in the same session. group 2 will be operated by cholecystectomy at least 6 months after bariatric surgery or whenever develop complications

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* presence of gallstone
* fit for laparoscopic surgery

Exclusion Criteria:

* BMI < 35
* unfit for surgery
* refuse to share in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
the incidence of complications | one year
  the incidence of complications of cholecystectomy or of left of gallstone

SECONDARY OUTCOMES:
operative time of cholecystectomy | 30-90 minutes
  operative time of cholecystectomy
%EWL | one year
  percentage of excess weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt